CLINICAL TRIAL: NCT02039921
Title: Observational, Retrospective, Multicenter Study to Describe the Reasons for the Change of Antiretroviral Treatment Regimen in HIV-positive Patients Between January 2011 and July 2012 in Spanish Hospitals
Brief Title: Observational, Retrospective, Multicenter Study to Describe the Reasons for the Change of the Regimen of Antiretroviral Therapy in HIV Patients
Acronym: SWITCHART
Status: Completed | Type: Observational
Sponsor: Fundacion SEIMC-GESIDA (Other)
Responsible Party: Sponsor
Other Study IDs: GESIDA-7913
Record Dates: First submitted 2014-01-15; First posted 2014-01-20 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2014-01

CONDITIONS: HIV

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study aims to describe the changes of combination antiretroviral therapy and the causes that motivated them.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients with HIV
* Patients in antiretroviral regimen, that have changed the antirretroviral treatment.

Exclusion Criteria:

* Patients unable to sign the consent form
* patients that changing their treatment are going to take the same components in co-formulated
* patients that changing their treatment are going to take the same components separately
* Total or selective interrupts not indicated by the specialist
* Patients that after changing antiretroviral therapy between January 2011 and July 2012, and during the next year, again suffered another change of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV patients that have changed antirretroviral régimen between Jan 2011 and Jul 2012
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of patients that change the treatment and the reason for it | 18 months
  Describe the changes in combination antiretroviral therapy and the causes that led, in patients with HIV infection, between January 2011 and July 2012 in routine clinical practice

CONTACTS AND LOCATIONS:
Locations (12):
- Spain (12):
  - Hospital Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Vall D'Hebron, Barcelona, Barcelona
  - Hospital San Cecilio, Granada, Granada
  - Hospital de Santiago de Compostela, Santiago de Compostela, La Coruña
  - Hospital Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Gregorio Marañón, Madrid, Madrid
  - Hospital La paz, Madrid, Madrid
  - Hospital Virgen de la Victoria, Málaga, Málaga
  - Hospital Virgen del Rocio, Seville, Sevilla
  - Hospital Miguel Servet, Zaragoza, Zaragoza